CLINICAL TRIAL: NCT03621397
Title: The Effectiveness of an Online Spanish Cognitive Intervention Program for Spanish-Speaking Latino/Hispanic Subarachnoid Hemorrhage Patients
Brief Title: Online Spanish Cognitive Intervention Program for Spanish-Speaking Latino/Hispanic Subarachnoid Hemorrhage Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We are no longer recruiting research participants for this study. Also, a co-investigator is no longer working at this institution and is no longer a part of this study.
Sponsor: DHR Health Institute for Research and Development (Other)
Responsible Party: Principal Investigator, Eduardo Estevis, Clinical Neuropsychologist, DHR Health Institute for Research and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1222300-1
Record Dates: First submitted 2018-07-31; First posted 2018-08-08 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Subarachnoid Hemorrhage; Cognitive Impairment; Quality of Life; Depression, Anxiety
Keywords: Spanish-speakers; Subarachnoid hemorrhage; Cognitive Intervention
MeSH Terms: conditions — Subarachnoid Hemorrhage; Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 40 Spanish-speaking research participants who have sustained a subarachnoid hemorrhage in the last 6 months will participate in the research study. Participants will be randomly assigned to one of two groups: 1) Cognitive intervention group (n = 20) or 2) Control group (n = 20). The Cognitive Intervention group will receive the cognitive intervention, while the Control group will not receive any intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Intervention Group (Experimental): Research participants in the cognitive intervention group will undergo a baseline neuropsychological evaluation. One week later, they will receive the online training program (brainHQ by Posit Science) three times a week for 45 minutes for a total of 12 weeks. This group will return one week after completing the online intervention program for their follow-up neuropsychological evaluation. They will then return again one year later for another follow-up neuropsychological evaluation.
  Interventions: Device: brainHQ by Posit Science
- Control Group (No Intervention): Research participants in the control group will undergo a baseline neuropsychological evaluation. They will then return 13 weeks after their baseline neuropsychological evaluation for a follow-up neuropsychological evaluation and again one year later.

INTERVENTIONS:
Device: brainHQ by Posit Science — This is an online cognitive training program. It consists of 29 online exercises that work out attention, brain speed, memory, people skills, navigation, and intelligence. The current study will focus on the following exercises: attention, brain speed (e.g., processing speed), executive function, and memory.
  Arms: Cognitive Intervention Group

SUMMARY:
The purpose of this research study is to examine the effectiveness of an online Spanish cognitive intervention program in Latino/Hispanic Spanish-speaking subarachnoid hemorrhage patients. In particular, the researchers will examine whether cognitive impairments associated with a subarachnoid hemorrhagic event improve after completing the online cognitive intervention program. Secondary outcomes of the research study include examining whether there is an improvement in research participants' quality of life and psychological functioning as a result of the online Spanish cognitive intervention program.

DETAILED DESCRIPTION:
40 Spanish-speaking research participants who have sustained a subarachnoid hemorrhage in the last 6 months will participate in the current research study. Participants will be randomly assigned to one of two groups: 1) Cognitive intervention group (n = 20) or 2) Control group (n = 20).

ELIGIBILITY:
Inclusion Criteria:

* History of a subarachnoid hemorrhage within the last 6-months. Must be confirmed by medical records and/or neurointerventionist radiologist
* 18 years and older
* Primarily Spanish-Speaking
* Able to read in Spanish
* Able to use a computer

Exclusion Criteria:

* History of neurological conditions (e.g., Alzheimer's disease, epilepsy, traumatic brain injury, brain tumor, encephalitis, meningitis, Parkinson's disease) other than subarachnoid hemorrhage
* History of neurodevelopment disorder (e.g., autism spectrum disorders, attention deficit-hyperactivity disorder)
* History of learning disabilities
* History of psychiatric illness (e.g., depression, anxiety, bipolar disorder, schizophrenia)
* Alcohol or illicit substance abuse or dependence
* Currently on medication(s) that may impact performance on the neuropsychological evaluation or online cognitive intervention program
* Severe expressive aphasia
* Upper extremities or vision problems that prevent participant from adequately using a computer or completing the neuropsychological evaluation
* Unable to commit to participate for the entire study including returning for one-year follow-up neuropsychological evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Spanish Rey Auditory Verbal Learning Test | 16 months
  This is a commonly used comprehensive verbal learning and memory test. The test consists of a 15-item word list that is presented five times. Participants are then asked to recall as many words following a brief delay and 20 minutes later. Raw scores from the following scales will be utilized: Total Recall, Short-Delayed Free Recall, Long-Delayed Free Recall, and Recognition Hits. Score values range from 0-to-15. These are considered participants' raw scores. Raw scores will then be converted to scaled scores based on available published normative data. All converted scores will be presented as scaled scores with a mean of ten and standard deviation of three in order to ensure that all scores are on a uniform scale. Scores falling at 1.5 standard deviations below the mean (scaled score ≤ 5) will be considered impaired. Scores that are above the 1.5 cut-off (scaled score ≥ 6) will be considered to be intact. Intact scores will be indicative of better memory outcomes.
Escala Wechsler de Inteligencia Para Adultos-IV (WAIS-IV; Wechsler, 2008) Retención de dígitos | 16 months
  This is an oral measure of working memory and attention abilities. Participants are presented with a series of numbers and must repeat them correctly in forward, reverse, and sequence order. Score values range from 0-to-48. These are considered participants' raw scores. Raw scores will then be converted to scaled scores based on available published normative data. All converted scores will be presented as scaled scores with a mean of ten and standard deviation of three in order to ensure that all scores are on a uniform scale. Scores falling at 1.5 standard deviations below the mean (scaled score ≤ 5) will be considered impaired. Scores that are above the 1.5 cut-off (scaled score ≥ 6) will be considered to be intact. Intact scores will be indicative of better outcomes on working memory and attentional abilities.
Escala Wechsler de Inteligencia Para Adultos-IV (WAIS-IV) Claves subtest | 16 months
  This is speeded graphomotor transcription subtest that assesses attention and processing speed abilities. Participants are required to a place a code with its designated number as quickly as possible in 120 seconds. Score values range from 0-to-135. These are considered participants' raw scores. Raw scores will then be converted to scaled scores based on available published normative data. All converted scores will be presented as scaled scores with a mean of ten and standard deviation of three in order to ensure that all scores are on a uniform scale. Scores falling at 1.5 standard deviations below the mean (scaled score ≤ 5) will be considered impaired. Scores that are above the 1.5 cut-off (scaled score ≥ 6) will be considered to be intact. Intact scores will be indicative of better outcomes on processing speed and attentional abilities.
Color Trails 1 and 2 (D'Elia, Satz, Lyons-Uchiyama, & White, 1996) | 16 months
  These two tests are non-verbal timed measures that assess processing speed and executive functioning abilities. Color Trails 1 is a sequencing test in which participants draw a line connecting numbers scattered throughout the test stimuli from least to greatest as quickly as possible. In Color Trails 2, participants are required to do the same as in Color Trails 1, but they must alternate colors for each number sequence as quickly as possible.
FAS (Lezak, 1995; Pontón et al., 1996; O'Bryant et al., 2017; Benton, Hamsher, & Sivan, 2000) | 16 months
  This is a measure of lexical fluency abilities. Participants are required to generate as many words as possible within 60 seconds with the letters F, A, and S.
Animal Naming (Lezak, 1995; O'Bryant et al., 2017 | 16 months
  This is a measure of semantic fluency abilities. Participants are required to generate as many animal names within 60 seconds.

SECONDARY OUTCOMES:
Spanish SF-36 (Ware, 1992; Alonso, 1995; Ware, 2000) | 16 months
  This is a 36-item quality of life measure. The 36-itmes are related to various aspects of the participants' life which are rated on a Likert scale of 1-to-5. From these items, the following eight subscales are derived: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role function, and mental. Scores on the SF-36 range from 1-100 with higher scores being indicative of better quality of life outcomes.
Spanish Satisfaction with Life Questionnaire (Diener, Emmons, Larsen, & Griffin, 1985; Diener & Gonzalez, 2011; Vásquez, Duque, & Hervás, 2013) | 16 months
  This is a 5-item questionnaire that assesses life satisfaction. These five items consist of Likert-scale responses that range from 1-7. Total scores on this measure range from 1-35 with higher scores being indicative of better life satisfaction outcomes.
Spanish Beck Depression Inventory-Second Edition (Beck, Steer, & Brown, 1996) | 16 months
  This is a 21-item depression self-report measure. These items consist of Likert-scale responses that range from 0-3 with lower scores being indicative of less depressive symptomology. Total scores range from 0-63. Cut-offs for depression severity is based on available published cut-off scores and includes the following ranges: minimal (0-13), mild (14-19), moderate (20-28), and severe (29-63). Participants who obtain classifications in the minimal range will be indicative of better psychological functioning outcomes. Participants who have scores in the moderate and severe range will be indicative of worse psychological functioning.
Spanish Beck Anxiety Inventory (Beck & Steer, 1993) | 16 months
  This is a 21-item anxiety self-report measure. These items consist of Likert-scale responses that range from 0-3 with lower scores being indicative of less anxiety. Total scores range from 0-63. Cut-offs for anxiety severity is based on available published cut-off scores and includes the following ranges: minimal (0-7), mild (8-15), moderate (16-25), and severe (26-63). Participants who obtain classifications in the minimal range will be indicative of better psychological functioning outcomes. Participants who have scores in the moderate and severe range will be indicative of worse psychological functioning.

OTHER OUTCOMES:
Spanish Marín Acculturation Scale (Marín et al., 1987) | One week
  This is a 13-item scale that assesses degree of acculturation. These items consist of 5-point Likert-scale responses with total scores ranging from 1-65. Low scores are suggestive of a low degree of acculturation and high scores are suggestive of a high degree of acculturation. This measure is not an outcome measure. It is use to establish level of acculturation. It will also be used in the data analysis to determine whether it impacts performance on cognitive measures.
Escala Wechsler de Inteligencia Para Adultos-IV (WAIS-IV) Vocabulario subtest | One week
  This is a Spanish oral measure of expressive vocabulary abilities. Participants are required to define words presented to them visually and orally. Score values range from 0-to-57. These are considered participants' raw scores. Raw scores will then be converted to scaled scores based on available published normative data. All converted scores will be presented as scaled scores with a mean of ten and standard deviation of three in order to ensure that all scores are on a uniform scale. Scores falling at 1.5 standard deviations below the mean (scaled score ≤ 5) will be considered impaired. Scores that are above the 1.5 cut-off (scaled score ≥ 6) will be considered to be intact. Intact scores will be indicative of participants' being Spanish-language dominant. This is not an outcome measure and only used to establish Spanish-language dominance.
Woodcock-Johnson III/Batería III Pruebas de aprovechamiento (Mather & Woodcock, 2005): Identificación de letras y palabras subtest: | One week
  This is a Spanish reading ability test. On this measure, participants are asked to name as many words as they can. This test initially begins with simple words and they increase in difficulty as the test progresses. Scores range from 1-76. These are considered participants' raw scores. Raw scores will then be converted to scaled scores based on available published normative data. All converted scores will be presented as scaled scores with a mean of ten and standard deviation of three in order to ensure that all scores are on a uniform scale. Scores falling at 1.5 standard deviations below the mean (scaled score ≤ 5) will be considered impaired. Scores that are above the 1.5 cut-off (scaled score ≥ 6) will be considered to be intact. Intact scores will be indicative of participants' being Spanish-language dominant. This is not an outcome measure and only used to establish Spanish-language dominance.
Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV; Wechsler, 2008) Vocabulary subtest | One week
  This is an English oral measure of expressive vocabulary abilities. Participants are required to define words presented to them visually and orally. Score values range from 0-to-57. These are considered participants' raw scores. Raw scores will then be converted to scaled scores based on available published normative data. All converted scores will be presented as scaled scores with a mean of ten and standard deviation of three in order to ensure that all scores are on a uniform scale. Scores falling at 1.5 standard deviations below the mean (scaled score ≤ 5) will be considered impaired. Scores that are above the 1.5 cut-off (scaled score ≥ 6) will be considered to be intact. Impaired scores will be indicative of participants' being Spanish-language dominant. This is not an outcome measure and is only being used to establish Spanish-language dominance.
Wide Range Achievement Test-Fourth Edition (WRAT-4; Wilkson & Robertson, 2006) Reading subtest | One week
  This is an English reading ability test. On this measure, participants are asked to name as many words as they can. This test initially begins with simple words and they increase in difficulty as the test progresses. Scores range from 0-70. These are considered participants' raw scores. Raw scores will then be converted to scaled scores based on available published normative data. All converted scores will be presented as scaled scores with a mean of ten and standard deviation of three in order to ensure that all scores are on a uniform scale. Scores falling at 1.5 standard deviations below the mean (scaled score ≤ 5) will be considered impaired. Scores that are above the 1.5 cut-off (scaled score ≥ 6) will be considered to be intact. Impaired scores will be indicative of participants' being Spanish-language dominant. This is not an outcome measure and is only being used to establish Spanish-language dominance.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Estevis, Ph.D., Principal Investigator — DHR Health
Locations (1):
- DHR Health Neuroscience Institute, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alonso J, Prieto L, Anto JM. [The Spanish version of the SF-36 Health Survey (the SF-36 health questionnaire): an instrument for measuring clinical results]. Med Clin (Barc). 1995 May 27;104(20):771-6. Spanish. PMID 7783470
- [Background] Beck, AT, Steer, RA. Beck Anxiety Inventory. San Antonio, TX: Psychological Corporation, 1993.
- [Background] Beck AT, Steer RA, Brown GK. Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation, 1996.
- [Background] Benton A L, Hamsher K, Sivan A. Multilingual Aphasia Examination: Manual. Iowa City, IA: AJA Associates Inc, 2000.
- [Background] brainHQ from Posit Science (https://es.brainhq.com/).
- [Background] D'Elia LF, Satz P, Lyons-Uchiyama C, White T. Color Trails Test Professional Manual. Lutz, FL: PAR, 1996.
- [Background] Lezak MD. Neuropsychological assessment (3rd ed.). New York, NY US: Oxford University Press, 1995.
- [Background] Marin G, Sabogal F, Otero-Sabogal R, Perez-Stable EJ. Development of a short acculturation scale for Hispanics. Hispanic Journal of Behavioral Sciences, 9, 183-205, 1987.
- [Background] Mather N, Woodcock RW. Manual de examinador (L.Wolfson, Trans). Woodcock-Johnson III Pruebas de aprovechamiento. Rolling Meadows, IL: Riverside, 2005.
- [Background] O'Bryant SE, Edwards M, Johnson L, Hall J, Gamboa A, O'jile J. Texas Mexican American adult normative studies: Normative data for commonly used clinical neuropsychological measures for English- and Spanish-speakers. Dev Neuropsychol. 2018 Jan;43(1):1-26. doi: 10.1080/87565641.2017.1401628. Epub 2017 Nov 30. PMID 29190120
- [Background] Ponton MO, Satz P, Herrera L, Ortiz F, Urrutia CP, Young R, D'Elia LF, Furst CJ, Namerow N. Normative data stratified by age and education for the Neuropsychological Screening Battery for Hispanics (NeSBHIS): Initial report. J Int Neuropsychol Soc. 1996 Mar;2(2):96-104. doi: 10.1017/s1355617700000941. PMID 9375194
- [Background] Rey A. L 'examen clinique en psychologie [Clinical tests in psychology]. Presses Universitaires de France, Paris, 1964.
- [Background] Schmidt M. Rey Auditory and Verbal Learning Test: a handbook. Los Angeles, CA: Western Psychological Services, 1996.
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Wechsler D. Wechsler Adult Intelligence Scale-Fourth Edition. San Antonio, TX: The Psychological Corporation, 2008.
- [Background] Wechsler D. Escala Wechsler de Inteligencia Para Adultos-IV. México D.F.: Editorial El Manual Moderno, NCS Pearson Inc, 2008.
- [Background] Wilkinson G, Robertson G. Wide range achievement test-fourth edition. Lutz, FL: Psychological Assessment Resources, Inc: 2006.
- [Result] Appelbaum PS, Grisso T. Assessing patients' capacities to consent to treatment. N Engl J Med. 1988 Dec 22;319(25):1635-8. doi: 10.1056/NEJM198812223192504. PMID 3200278
- [Result] Barnes DE, Yaffe K, Belfor N, Jagust WJ, DeCarli C, Reed BR, Kramer JH. Computer-based cognitive training for mild cognitive impairment: results from a pilot randomized, controlled trial. Alzheimer Dis Assoc Disord. 2009 Jul-Sep;23(3):205-10. doi: 10.1097/WAD.0b013e31819c6137. PMID 19812460
- [Result] Dreer LE, Devivo MJ, Novack TA, Krzywanski S, Marson DC. Cognitive Predictors of Medical Decision-Making Capacity in Traumatic Brain Injury. Rehabil Psychol. 2008 Nov 1;53(4):486-497. doi: 10.1037/a0013798. PMID 20686627
- [Result] Egeto P, Loch Macdonald R, Ornstein TJ, Schweizer TA. Neuropsychological function after endovascular and neurosurgical treatment of subarachnoid hemorrhage: a systematic review and meta-analysis. J Neurosurg. 2018 Mar;128(3):768-776. doi: 10.3171/2016.11.JNS162055. Epub 2017 Apr 14. PMID 28409729
- [Result] Estevis E, Basso MR, Combs D. Effects of practice on the Wechsler Adult Intelligence Scale-IV across 3- and 6-month intervals. Clin Neuropsychol. 2012;26(2):239-54. doi: 10.1080/13854046.2012.659219. Epub 2012 Feb 21. PMID 22353021
- [Result] Fernandez-Calvo B, Rodriguez-Perez R, Contador I, Rubio-Santorum A, Ramos F. [Efficacy of cognitive training programs based on new software technologies in patients with Alzheimer-type dementia]. Psicothema. 2011 Feb;23(1):44-50. Spanish. PMID 21266141
- [Result] Kesler S, Hadi Hosseini SM, Heckler C, Janelsins M, Palesh O, Mustian K, Morrow G. Cognitive training for improving executive function in chemotherapy-treated breast cancer survivors. Clin Breast Cancer. 2013 Aug;13(4):299-306. doi: 10.1016/j.clbc.2013.02.004. Epub 2013 May 4. PMID 23647804
- [Result] Latimer SF, Wilson FC, McCusker CG, Caldwell SB, Rennie I. Subarachnoid haemorrhage (SAH): long-term cognitive outcome in patients treated with surgical clipping or endovascular coiling. Disabil Rehabil. 2013 May;35(10):845-50. doi: 10.3109/09638288.2012.709909. Epub 2012 Aug 22. PMID 22909316
- [Result] Marson DC, Strickland A, Hethcox A, DeVivo M, Taylor S, Krzywanski S, et al. Assessing competency to consent to treatment in traumatic brain injury. Paper presented at the 21st Annual Conference of the National Academy of Neuropsychology, San Francisco, California, 2001.
- [Result] Penner IK, Vogt A, Stocklin M, Gschwind L, Opwis K, Calabrese P. Computerised working memory training in healthy adults: a comparison of two different training schedules. Neuropsychol Rehabil. 2012;22(5):716-33. doi: 10.1080/09602011.2012.686883. Epub 2012 Jun 6. PMID 22671966
- [Result] Westerberg H, Jacobaeus H, Hirvikoski T, Clevberger P, Ostensson ML, Bartfai A, Klingberg T. Computerized working memory training after stroke--a pilot study. Brain Inj. 2007 Jan;21(1):21-9. doi: 10.1080/02699050601148726. PMID 17364516